CLINICAL TRIAL: NCT02697630
Title: A Multicenter Phase II Open Label Study to Evaluate Efficacy of Concomitant Use of Pembrolizumab and Entinostat in Adult Patients With Metastatic Uveal Melanoma
Brief Title: Efficacy Study of Pembrolizumab With Entinostat to Treat Metastatic Melanoma of the Eye
Acronym: PEMDAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1
Record Dates: First submitted 2016-02-22; First posted 2016-03-03 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Uveal Melanoma
Keywords: Uveal melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — pembrolizumab; entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Entinostat (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Entinostat

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg administered intravenously (IV) every third week until progression or unacceptable toxicity for a maximum of 24 months
Drug: Entinostat — 5 mg by mouth (PO) once weekly until progression or unacceptable toxicity for a maximum of 24 months

SUMMARY:
The purpose of this study is to see if the combination of entinostat and pembrolizumab can be an effective treatment for patients with melanoma of the eye (uveal melanoma) that has spread to other sites of the body (metastatic disease). Pembrolizumab is an antibody that helps the immune system to attack cancer cells. Although pembrolizumab has proven clinical efficacy in treating patients with metastatic cutaneous melanoma, an effect on metastatic uveal melanoma has not been established. Entinostat is a histone deacetylase (HDAC) inhibitor that has effects on both cancer cells and immune regulatory cells, thus potentially enhancing the effects of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Signed and dated written informed consent before the start of specific protocol procedures.
* ECOG PS 0-1
* Histologically/cytologically confirmed stage IV uveal melanoma
* Measurable disease by computed tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST 1.1 criteria
* Any number of prior therapies (including none), with the exception of anticancer immunotherapy

Exclusion Criteria:

* Active brain metastases (symptomatic and/or requiring corticosteroids) or leptomeningeal metastases
* Previous treatment with anticancer immunotherapy
* Pregnant or nursing (lactating) women
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study
* Active autoimmune disease
* Immune deficiency or treatment with systemic corticosteroids
* Use of other investigational drugs (drugs not marketed for any indication) within 28 days before study drug administration
* Life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From first dose up to 24 months
  The proportion of patients that have a best overall response of complete response (CR) or partial response (PR), as assessed by RECIST 1.1.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | 18 weeks from first dose
Progression free survival (PFS) | From first dose up to 24 months
Overall Survival (OS) | From first dose up to 24 months
Best overall response (BOR) | From first dose up to 24 months
Time To Response (TTR) | From first dose up to 24 months
Duration of objective response (DOR) | From first dose up to 24 months
Adverse Events (AEs) and Serious Adverse Events (SAEs). | From first dose up to 24 months
  Incidence and severity
Eastern Cooperative Oncology Group (ECOG) Performance status (PS) | 18 weeks from first dose
Quality of Life (QoL) assessed by FACT-G | From first dose up to 24 months
Quality of Life (QoL) assessed by EQ5D-3L | From first dose up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of oncology, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ny L, Jespersen H, Karlsson J, Alsen S, Filges S, All-Eriksson C, Andersson B, Carneiro A, Helgadottir H, Levin M, Ljuslinder I, Olofsson Bagge R, Sah VR, Stierner U, Stahlberg A, Ullenhag G, Nilsson LM, Nilsson JA. The PEMDAC phase 2 study of pembrolizumab and entinostat in patients with metastatic uveal melanoma. Nat Commun. 2021 Aug 27;12(1):5155. doi: 10.1038/s41467-021-25332-w. PMID 34453044
- [Result] Sah VR, Jespersen H, Karlsson J, Nilsson LM, Bergqvist M, Johansson I, Carneiro A, Helgadottir H, Levin M, Ullenhag G, Stahlberg A, Olofsson Bagge R, Nilsson JA, Ny L. Chemokine Analysis in Patients with Metastatic Uveal Melanoma Suggests a Role for CCL21 Signaling in Combined Epigenetic Therapy and Checkpoint Immunotherapy. Cancer Res Commun. 2023 May 18;3(5):884-895. doi: 10.1158/2767-9764.CRC-22-0490. eCollection 2023 May. PMID 37377898
- [Result] Jespersen H, Olofsson Bagge R, Ullenhag G, Carneiro A, Helgadottir H, Ljuslinder I, Levin M, All-Eriksson C, Andersson B, Stierner U, Nilsson LM, Nilsson JA, Ny L. Concomitant use of pembrolizumab and entinostat in adult patients with metastatic uveal melanoma (PEMDAC study): protocol for a multicenter phase II open label study. BMC Cancer. 2019 May 2;19(1):415. doi: 10.1186/s12885-019-5623-3. PMID 31046743